CLINICAL TRIAL: NCT06319755
Title: Characteristics of Intestinal Microbiome Following Pancreatic Surgery - a Prospective Case Controlled Exploratory Study
Brief Title: Characteristics of Intestinal Microbiome Following Pancreatic Surgery
Status: Recruiting | Type: Observational
Sponsor: Royal Prince Alfred Hospital, Sydney, Australia (Other)
Responsible Party: Principal Investigator, Dale Palmer, Clinical Dietitian, Royal Prince Alfred Hospital, Sydney, Australia
Other Study IDs: X23-0230
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Cancer; Microbiota; Pancreatoduodenectomy
Keywords: matched case control study
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Post-surgical patients: Adults having had pancreatoduodenectomy (Whipple's) surgery for curative intent.
- Matched controls: Participants matched to each post-surgical participant by age, sex, body mass index (BMI), smoking status.

SUMMARY:
The goal of this observational study is to learn about intestinal microbiome structure and function in individuals who have undergone a pancreatoduodenectomy and compare to healthy matched controls.

The primary objectives of the study are:

1. To explore and describe any differences in the gut microbiota especially Shannon diversity index
2. To conduct functional profiling by exploring and describing any differences in functional metabolites produced in the gut in people having had pancreatoduodenectomy greater than 6 months ago compared to healthy matched controls.

Participants will be asked to complete the following:

* Three-day food, bowel and medication diary (see Protocol appendix 5)
* Gastrointestinal Symptom Rating Scale (see Protocol appendix 6)
* Quality of life questionnaire (see Protocol appendix 7)
* Stool sample test using Microba Insight TradeMark (a small swab is taken from soiled toilet paper, sealed in a room-temperature storage capsule and mailed to the testing laboratory)

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged equal to or greater than 18 years) having had pancreatoduodenectomy (Whipple's) surgery between April 2018 - December 2023 for curative intent and received post-operative clinical management at Royal Prince Alfred Hospital, (post-surgical participants), and
* Healthy adults matched by age, sex, body mass index and smoking status

Exclusion Criteria:

* Aged less than 18 years
* Are unable to complete the questionnaires or testing due to language or cognitive limitations
* Have active or recurring pancreatic cancer, or where the surgery was for non-curative intent
* Have other gastrointestinal conditions that could affect gut symptoms or microbiome such as Inflammatory Bowel disease, Irritable Bowel Syndrome Coeliac disease, or are currently pregnant or breastfeeding
* Are currently taking medications or diet that can affect gut symptoms or microbiome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post-surgical patients are adults (aged ≥ 18 years) who have undergone a pancreatoduodenectomy (Whipple's) surgery for curative between the time period of April 2018 - December 2023, and received post-operative clinical management at Royal Prince Alfred Hospital. Healthy adults (matched controls) will be matched by age, sex, body mass index and smoking status.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of microbiota profile between post-surgical participants and healthy controls. | During data collection, 3 days
  Stool samples will be analysed to compare the Shannon diversity index (calculated by taking the number of each microbial species, the proportion each species is of the total number of individuals, summed by the proportion times the natural log of the proportion for each species) between participant groups.

SECONDARY OUTCOMES:
Compliance with 3-day food dairies | From enrollment to the collection of data from participants, 3 days
  Compliance with 3-day food dairies (completion rate of food diaries)
Pre-paid return rates | From enrollment to the collection of data from participants, 3 days
  Pre-paid return rates (proportion (number) of envelopes returned)
Ease of matching | Enrollment period, up to 12 months
  Ease of matching (ability to match surgical patients to controls based on age, gender, body mass index, smoking status)
Shannon diversity index | During data collection period, 3 days
  Shannon diversity index (calculated by taking the number of each microbial species, the proportion each species is of the total number of individuals, summed by the proportion times the natural log of the proportion for each species)
Gastrointestinal symptoms | During data collection period, 3 days
  Gastrointestinal symptoms (total number of bowel motions)
Protein:fibre ratio of diet | During data collection period, 3 days
  Protein:fibre ratio of diet (average grams of protein consumed divided by grams of fibre consumed)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition and Dietetics, Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No